CLINICAL TRIAL: NCT03247985
Title: Randomized Prospective Single-Blinded Study of Totally Extra Peritoneal Inguinal Hernia Repair: Tacking Mesh Versus Self-fixating Mesh
Brief Title: Tacking Mesh Versus Self-fixating Mesh for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David R. Farley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-003616
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Results first posted 2017-11-17 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Hernia, Inguinal
Keywords: Mesh; Repair; Peritoneal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PROLENE Polypropylene Tacking Mesh (Active Comparator): Participants will be randomized to Tacking Mesh for their inguinal hernia surgery.
  Interventions: Device: PROLENE Polypropylene Tacking Mesh
- ProGrip Self-fixating Mesh (Active Comparator): Participants will be randomized to Self-fixing mesh for their inguinal hernia surgery
  Interventions: Device: ProGrip Self-fixating Mesh

INTERVENTIONS:
Device: PROLENE Polypropylene Tacking Mesh — Prolene mesh is a polypropylene plastic mesh (10 x 15 cm) implant fixed with titanium tacks
  Arms: PROLENE Polypropylene Tacking Mesh
Device: ProGrip Self-fixating Mesh — ProGrip™ self-fixating mesh is a tack-free fixation mesh for use in open & laparoscopic hernia repairs. It is composed of absorbable Monofilament Polylactic Acid micro grips on one surface integrated with a lightweight Monofilament Polyethylene Terephthalate. The micro grips act as a kind of "Velcro" to the soft tissue surfaces resulting in self-fixation
  Arms: ProGrip Self-fixating Mesh

SUMMARY:
Investigators are testing whether tacking mesh or self-fixating mesh used for inguinal hernia repair makes any difference in short-term pain or return to normal activities following the operation. Other studies have shown no significant difference in hernia recurrence rate when metal tacks are not used to hold the mesh in place.

DETAILED DESCRIPTION:
Participants will be placed into two groups. One group of participants will have mesh tacked into place for their hernia repairs. The other group will have self-fixating mesh into place. Both groups will have a piece of mesh that will widely cover the hernia defect. Before surgery, the participant will be asked to rate discomfort on a 0-10 scale. Zero stands for no pain and 10 is the worst pain they can imagine. Investigators will record information about general medical condition, medications and activity level. During the operation information will be recorded about the pain medicines the participant may receive. In the recovery room the participant will be asked to rate their pain on the 0-10 scale and more information will be recorded about any additional pain medicines that they may receive and assess activity level. Following surgery, Investigators will contact the participants by survey to obtain more information about pain level, medication use, and activity level.

ELIGIBILITY:
Inclusion Criteria:

- All patients regardless of sex or age who were diagnosed with a inguinal hernia and underwent a totally extraperitoneal (TEP) inguinal hernia repair at the Mayo Clinic in Rochester, Minnesota from June 2013 - June 2014.

Exclusion Criteria:

- Patients who did not elect to undergo a hernia repair or who elected to undergo a different type of hernia repair instead of a TEP procedure.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Farley, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Mayo Clinic in Rochester, Minnesota from June 2013 to June 2014.
Period: Overall Study
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11) | 55 (11) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 19 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30 (10) | 30 (4) | 30 (9)
Site of Hernia [Count of Participants; unit: Participants]
  Unilateral | 3 | 8 | 11
  Bilateral | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Operative Time
Description: Length of time needed to complete surgery.
Time Frame: First incision to closure, approximately one hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
Number analyzed (Participants) | 19 | 19
minutes
  Bilateral | 69 (6.5) | 84 (7.8)
  Unilateral | 40 (12) | 66 (7)
Statistical Analysis 1: Comparison: PROLENE Polypropylene Tacking Mesh vs ProGrip Self-fixating Mesh; Comparison between groups for bilateral operative time; Test type: Superiority; p = 0.17, t-test, 2 sided
Statistical Analysis 2: Comparison: PROLENE Polypropylene Tacking Mesh vs ProGrip Self-fixating Mesh; Comparison between groups for unilateral operative time; Test type: Superiority; p = 0.09, t-test, 2 sided

2. Primary Outcome: Number of Participants With Early Postoperative Complications
Description: Any complication which occurred within 30 days after the operation.
Time Frame: Within 30 days
Measure: Number; unit: participants
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
Number analyzed (Participants) | 19 | 19
participants
  Overnight admittance to hospital | 2 | 1
  Urinary retention | 1 | 1
  Skin infection | 1 | 0
  Recurrence of hernia | 0 | 1

3. Secondary Outcome: Pain Score at Baseline
Description: Participants were asked to rate their level of pain on a Likert scale (0 through 5; 0=no pain, 5=severe pain).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
Number analyzed (Participants) | 19 | 19
units on a scale | 1.13 (1.196) | 1.5 (1.29)

4. Secondary Outcome: Pain Score at One Week
Description: Participants were asked to rate their level of pain on a Likert scale (0 through 5; 0=no pain, 5=severe pain).
Time Frame: One Week Postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
Number analyzed (Participants) | 19 | 19
units on a scale | 1.1 (0.904) | 0.8 (0.747)
Statistical Analysis 1: Comparison: PROLENE Polypropylene Tacking Mesh vs ProGrip Self-fixating Mesh; A p-value of 0.05 was considered statistically significant; Test type: Superiority; p = 0.02, t-test, 2 sided

5. Secondary Outcome: Pain Score at Four Weeks
Description: Participants were asked to rate their level of pain on a Likert scale (0 through 5; 0=no pain, 5=severe pain).
Time Frame: Four Weeks Postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
Number analyzed (Participants) | 19 | 19
units on a scale | 0.1 (0.236) | 0.3 (0.757)

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | PROLENE Polypropylene Tacking Mesh | ProGrip Self-fixating Mesh
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/19
Other Adverse Events (participants affected / at risk) | 1/19 | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROLENE Polypropylene Tacking Mesh (N=19) | ProGrip Self-fixating Mesh (N=19)
Admission to hospital (Renal and urinary disorders) | 2 (2) | 1 (1) — Bladder catheterization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROLENE Polypropylene Tacking Mesh (N=19) | ProGrip Self-fixating Mesh (N=19)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Inguinal Hernia Recurrence (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The small sample size limits the power to reflect statistical differences. This study had a large number of bilateral repairs reflecting the inherent referral bias of our practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes